CLINICAL TRIAL: NCT07070817
Title: A Clinical Study of Ultrasound-guided Botulinum Toxin A Into Salivary Gland for Sialorrhea After True Bulbar Palsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: houyajing (Other)
Responsible Party: Sponsor-Investigator, houyajing, Fuxing Hospital affiliated to Capital Medical University, Fu Xing Hospital, Capital Medical University
Organization: Fu Xing Hospital, Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024FXHEC-KSP017
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Sialorrhea True Bulbar Palsy Medullary Injury
MeSH Terms: interventions — incobotulinumtoxinA; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, double-blind interventional study designed to evaluate the efficacy and safety of ultrasound-guided botulinum toxin type A (BTX-A) injection into salivary glands for treating sialorrhea in patients with true bulbar palsy. The study adopts a parallel-group design with a 1:1 allocation ratio between the experimental group and the control group, following strict randomization and blinding procedures to ensure the objectivity and reliability of results.
  1.Study Design Type
  A randomized controlled trial (RCT) with a parallel-group design, comparing two intervention strategies:
  1.1Control group (Group A): Routine swallowing rehabilitation training. 1.2Experimental group (Group B): Ultrasound-guided BTX-A injection into the parotid and submandibular glands, combined with the same routine swallowing rehabilitation training as the control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Use a randomization tool to generate a random number table and set a seed number. Generate random envelopes based on the random code table. Cases that meet the inclusion and exclusion criteria will be enrolled in sequence according to the content of the random envelopes in the order of enrollment. Researchers responsible for enrolling patients will recruit patients. Those assigned to the botulinum toxin group will receive type A botulinum toxin (diluted with 2ml of 0.9% NaCl) plus routine swallowing rehabilitation training."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Botulinum Toxin Type A (BoNT-A) Salivary Gland Injection Group (Experimental): Experimental Arm (Group B) Intervention: Participants receive ultrasound-guided A 100IU (BTX-A) injection into the salivary glands combined with the same routine swallowing rehabilitation training as the control arm.
  Details of BTX-A injection:
  BTX-A is diluted with 2 mL of 0.9% NaCl. Injections are administered under ultrasound guidance, targeting the parotid and submandibular glands (specific dosage and injection sites follow clinical standards).
  Rehabilitation training: Identical in content, frequency, and duration to the control arm, ensuring that any differences in outcomes can be attributed to the BTX-A injection.
  Interventions: Drug: Ultrasound-Guided Botulinum Toxin Type A (BoNT-A) Salivary Gland Injection
- Ultrasound-Guided Saline (Placebo) Salivary Gland Injection Group (Placebo Comparator): Description: This arm includes participants with true bulbar palsy and sialorrhea who will receive ultrasound-guided injections of a placebo (sterile saline) into the salivary glands. It serves as a control to compare against the active intervention arm.
  Interventions: Drug: Control (Normal saline)

INTERVENTIONS:
Drug: Ultrasound-Guided Botulinum Toxin Type A (BoNT-A) Salivary Gland Injection — Ultrasound-guided injection of BoNT-A (specific dosage, e.g., "100 units") into target salivary glands ( parotid and submandibular glands) at baseline.
  Arms: Ultrasound-Guided Botulinum Toxin Type A (BoNT-A) Salivary Gland Injection Group
Drug: Control (Normal saline) — Intervention: Participants receive routine swallowing rehabilitation training only.
  Details of training: The training includes standard techniques to improve swallowing function, such as oral motor training, empty swallowing exercises, and ice stimulation. The frequency and duration of training are consistent across all participants in this arm to ensure standardization.
  Arms: Ultrasound-Guided Saline (Placebo) Salivary Gland Injection Group

SUMMARY:
Sialorrhea refers to a group of syndromes characterized by excessive saliva secretion from the salivary glands or reduced clearance of oral saliva due to dysphagia, resulting in saliva overflowing from the corners of the mouth or accumulating in the pharynx. It is one of the common clinical problems in conditions such as cerebral palsy, Parkinson's disease [1], and brain injuries (including stroke, traumatic brain injury, and hypoxic-ischemic encephalopathy). Among them, true bulbar palsy after medullary injury often causes saliva to flow out from the corners of the mouth due to sensory impairment in the oral cavity, tongue, and pharynx, as well as motor dysfunction and loss of coordination of swallowing-related muscles [2]; on the other hand, it often leads to residual saliva in the hypopharynx due to weakness of the pharyngeal constrictor muscles and dysfunction of the upper esophageal sphincter [3]. Sialorrhea can not only cause oral odor, skin breakdown, and malnutrition but also have a negative impact on patients' psychology, and even lead to choking or aspiration pneumonia, seriously endangering their physical and mental health. Therefore, active management and treatment of sialorrhea in patients with true bulbar palsy have become the key to solving this problem.

Currently, the management of sialorrhea mainly involves improving swallowing function to enhance saliva clearance and using drug intervention to reduce saliva secretion, thereby alleviating sialorrhea symptoms. However, current studies have found that swallowing function cannot recover quickly in a short time in patients with medullary injury. Therefore, active intervention is needed to reduce saliva secretion to relieve sialorrhea symptoms. Clinical treatments for sialorrhea include drug therapy, botulinum toxin therapy, radiation therapy, and surgical treatment. Among them, oral drug therapy is mainly based on antimuscarinic drugs. Although it has a certain therapeutic effect, its clinical application is limited due to the side effects of systemic anticholinergic effects; while surgical treatment is not clinically adopted because of its high destructiveness.

In recent years, a number of clinical studies on botulinum toxin type A (BTX-A) in the treatment of sialorrhea in adults (Parkinson's disease, traumatic brain injury) and children (cerebral palsy) have been carried out at home and abroad, and its efficacy and safety have been verified [4] [5]. However, there are few reports on BTX-A in the treatment of sialorrhea in patients with medullary lesions. Therefore, this study aims to conduct a randomized controlled trial to explore the effect of ultrasound-guided botulinum toxin type A injection into the salivary glands on sialorrhea in patients with true bulbar palsy, and comprehensively evaluate the efficacy and safety of BTX-A in the treatment of sialorrhea by combining subjective scale assessment and objective instrument assessment.

ELIGIBILITY:
Inclusion Criteria:① Aged 18-80 years; ② Cerebral magnetic resonance imaging or computed tomography confirms medullary lesions (hemorrhage, ischemia, or tumor); ③ Dysphagia is clearly diagnosed by flexible endoscopic evaluation of swallowing (FEES); ④ Presence of sialorrhea, which is defined as meeting any one of the following three criteria: total score of the Drooling Severity and Frequency Scale (DSFS-T) ≥ 4 points, each item score of the Drooling Severity and Frequency Scale (DSFS) ≥ 2 points, or score of the Murray Secretion Scale (MSS) for pharyngeal secretions ≥ 2 points; ⑤ Conscious and able to cooperate with sialorrhea assessment and follow-up; ⑥ Willing to receive BTX-A injection, informed of the study details, and sign the relevant informed consent documents.

-

Exclusion Criteria:① Having received BTX-A injection treatment in the recent six months;

* Having an allergy or contraindication to botulinum toxin;

  * Having taken drugs for treating sialorrhea or drugs that can cause sialorrhea in the recent month;

    * Having severe diseases of important organs such as the heart, lungs, liver, kidneys, or malignant tumors, etc.; ⑤ Concomitantly using aminoglycoside antibiotics and warfarin; ⑥ Patients with infection or skin lesions at the injection site, or severe muscle atrophy at the injection site, or those with infection at the injection site, or skin lesions at the injection site, or severe muscle atrophy at the injection site, or infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Global Impression of Change Scale (GICS) assessment: | The Global Impression of Change Scale (GICS) will be used to assess symptoms at 1 week, 2 weeks, and 4 weeks after injection treatment.
  This scale rates the patient's current condition by comparing it with the initial condition, with scores ranging from 0 to 7. The specific criteria are as follows:
  This scale rates the patient's current condition by comparing it with the initial condition, with scores ranging from 0 to 7. The specific criteria are as follows:
  0 points: Not evaluated
  1. point: Significant improvement
  2. points: Improvement
  3. points: Slight improvement
  4. points: No change
  5. points: Slight deterioration
  6. points: Deterioration
  7. points: Severe deterioration

SECONDARY OUTCOMES:
Flexible Endoscopic Evaluation of Swallowing (FEES) combined with Murray Secretion Scale (MSS) assessment: | Murray Secretion Scale (MSS) will be used to assess the patients' sialorrhea symptoms before BTX-A treatment, as well as 1 week, 2 weeks, and 4 weeks after treatment, respectively.
  A flexible laryngoscope is inserted through one nostril to observe the retention of secretions in the vallecula epiglottica, piriform fossa, and laryngeal vestibule, and the MSS is used for scoring. The scoring criteria are as follows:
  0 points: No secretions in the vallecula epiglottica and piriform fossa
  1. point: A small amount of secretions in the vallecula epiglottica and piriform fossa
  2. points: Temporary accumulation of secretions in the laryngeal vestibule
  3. points: Persistent accumulation of secretions in the laryngeal vestibule
Assessment with Drooling Severity and Frequency Scale (DSFS) | The Drooling Severity Scale (DSFS-S), Drooling Frequency Scale (DSFS-F) will be used to assess the patients' sialorrhea symptoms before BTX-A treatment, as well as 1 week, 2 weeks, and 4 weeks after treatment, respectively.
  Drooling Severity Scale (DSFS-S): The score ranges from 1 to 5, with 1 point indicating normal; 2 points indicating mild (only the lips are moist); 3 points indicating moderate (the mouth and chin are moist); 4 points indicating severe (clothes are damp); 5 points indicating persistent drooling (clothes, hands and surrounding objects are moist).
  Drooling Frequency Scale (DSFS-F): The score ranges from 1 to 5, with 1 point indicating no drooling; 2 points indicating occasional drooling (not every day); 3 points indicating frequent drooling (some time every day); 4 points indicating constant drooling.
  The total score of the overall scale is the sum of the scores of the two subscales, ranging from 2 to 9 points. A score of 2 indicates no drooling, and a score of 9 indicates severe drooling. A higher score suggests a more severe degree of drooling.
Assessment with Hamilton Anxiety Scale | The incidence of depression in the two groups of patients will be compared before BTX-A treatment and2weeks and 4 weeks a after treatment.
  All items are evaluated using a 5-level scoring method with scores ranging from 0 to 4: 0 points indicate no symptoms; 1 point indicates mild symptoms; 2 points indicate moderate symptoms; 3 points indicate severe symptoms; 4 points indicate extremely severe symptoms.
  A total score of <7 points indicates no anxiety, 7-13 points indicates possible anxiety, 14-20 points indicates anxiety, 21-28 points indicates obvious anxiety, and ≥29 points indicates severe anxiety. Among them, a score of ≥14 points suggests that the evaluated person has clinically significant anxiety symptoms.
Assessment with Hamilton Depression Scale | The incidence of Anxiety in the two groups of patients will be compared before BTX-A treatment and 2weeks and 4 weeks after treatment.
  Most items are evaluated using a 5-level scoring method with scores ranging from 0 to 4 (0 points indicate no symptoms; 1 point indicates mild symptoms; 2 points indicate moderate symptoms; 3 points indicate severe symptoms; 4 points indicate extremely severe symptoms); a few items are evaluated using a 3-level scoring method with scores ranging from 0 to 2 (0 points indicate no symptoms; 1 point indicates mild to moderate symptoms; 2 points indicate severe symptoms).
  A total score of <8 points indicates no depression, 8-19 points indicates possible depression, 20-34 points indicates mild or moderate depression, and ≥35 points indicates severe depression. Among them, a score of ≥20 points suggests that the patient has clinically significant depressive symptoms.
Occurrence of Pulmonary Infection | The incidence of stroke-associated pneumonia in the two groups of patients will be compared before BTX-A treatment and 2 weeks after treatment.
  It is judged according to the diagnostic criteria for stroke-associated pneumonia, that is, chest imaging examination reveals new or progressive pulmonary infiltrative lesions, accompanied by more than 2 clinical infection symptoms (such as fever > 38℃; new onset of cough and expectoration or aggravation of original respiratory disease symptoms, with dyspnea or tachypnea, respiratory rate > 25 times/min; signs of pulmonary consolidation and/or rales; peripheral blood leukocytes > 10.0×10⁹/L or < 4.0×10⁹/L, excluding interstitial lung changes, pulmonary edema, atelectasis, and pulmonary embolism); or age ≥ 70 years old with altered consciousness for no other clear reasons.
The main indicators include prealbumin, serum albumin (Alb), and hemoglobin (Hb). | The improvement of nutritional status in the two groups of patients will be compared before BTX-A treatment and 2 weeks after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuxing Hospital Affiliated to Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No